CLINICAL TRIAL: NCT03171428
Title: Hepatectomy With or Without the Thoraco-abdominal Approach: Impact on Perioperative Outcome
Brief Title: Hepatectomy With or Without the Thoraco-abdominal Approach
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Prof. Guido Torzilli, Director of the Department of Hepatobiliary Surgery, University of Milan
Other Study IDs: ThoraxForLiver
Record Dates: First submitted 2017-05-28; First posted 2017-05-31 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Surgery; Liver Tumors; Hepatectomy; Liver Resection
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TAA: Thoraco-Abdominal Approach: those patients with liver tumors operated with the thoracic-abdominal approach
  Interventions: Procedure: Hepatectomy
- AA: Abdominal Approach: those patients with liver tumors operated with the abdominal approach (without the thoracotomy)
  Interventions: Procedure: Hepatectomy

INTERVENTIONS:
Procedure: Hepatectomy — Surgery for liver tumors is the removal of a part of the liver affected by a tumor.
  Other Names: hepatic resection; liver resection; liver surgery

SUMMARY:
The performance of hepatectomy for liver tumors using the thoraco-abdominal approach (TAA) versus the abdominal approach (AA) is still debated.

The aim of the study is the analysis of the perioperative outcome of patients operated with or without the TAA for liver tumors.

DETAILED DESCRIPTION:
The prospectively maintained database was queried. A 1:1 propensity score-matched analysis was applied. Among 744 patients, 246 undergoing hepatectomy with TAA and 246 undergoing hepatectomy with AA were compared. These patients were matched for baseline characteristics, underlying liver disease, comorbidity, tumor features, and extent of the resection. The rates of morbidity and mortality were the study endpoints.

ELIGIBILITY:
Inclusion Criteria:

* First liver surgery;
* Any type of malignant liver tumor, including hepatocellular carcinoma on cirrhosis.

Exclusion Criteria:

* Previous history of liver surgery;
* Any type of benign liver tumor;
* Incomplete clinical, surgical, pathological or postoperative data;
* Patients treated with radiofrequency ablation alone or in combination with surgery were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by liver tumors scheduled for hepatectomy at our center.
Sampling Method: Probability Sample
Enrollment: 744 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2015-04-01 (Actual)

PRIMARY OUTCOMES:
Short-term outcome: Occurrence of postoperative complications or death after surgery | Within 90-days after the operation
  Occurrence of postoperative complications or death after surgery

IPD SHARING:
Plan to Share IPD: No